CLINICAL TRIAL: NCT07016659
Title: Assessing Antiplaque And Antigingivitis Efficacy Of Triphala Mouthwash Versus Chlorhexidine Mouthwash Among A Group Of Children: A Randomized Clinical Trial
Brief Title: Triphila Mouthwash Effect as Anti-plaque and Anti-gingivitis in Children
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Emad Abdelrazik Ahmed, Pediatric Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Triphila as antiplaque
Record Dates: First submitted 2025-05-29; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Plaque Accumulation; Gingival Inflammation
Keywords: triphila mouthwash; anti-plaque; anti-gingivitis; children
MeSH Terms: conditions — Gingivitis | interventions — hexitol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- use 0.12% Chlorhexidine mouthwash to asses its anti-plaque and anti-gingivitis effect (Placebo Comparator)
  Interventions: Drug: 0.12% Chlorhexidine Mouthwash ( Hexitol )
- use Triphala mouthwash to asses its anti-plaque and anti-gingivitis effect (Experimental)
  Interventions: Drug: Triphila mouthwash

INTERVENTIONS:
Drug: 0.12% Chlorhexidine Mouthwash ( Hexitol ) — About 10 ml will be administered, and participants will be asked to swish mouthwash for 30 seconds two times daily under the supervision of their parents, 30 to 45 minutes after toothbrushing for 2 weeks.
  Arms: use 0.12% Chlorhexidine mouthwash to asses its anti-plaque and anti-gingivitis effect
Drug: Triphila mouthwash — The participant will be instructed to administer 15 ml of the mouthwash and swish it for 30 seconds two times daily under the supervision of their parents, 30 to 45 minutes after toothbrushing for 2 weeks
  Arms: use Triphala mouthwash to asses its anti-plaque and anti-gingivitis effect

SUMMARY:
The study aim to to assess the antiplaque and antigingivitis efficacy of Triphala mouthwash versus chlorhexidine mouthwash among children.

Oral health, acknowledged as equally significant to general health, has become an essential component of an individual's entire well-being. Dental caries and periodontal problems are the two predominant oral conditions that repeatedly affect nearly all individuals throughout their entire lives (Sharma et al., 2014).

Numerous bacterial communities can be found in the oral cavity. These bacteria are harmless if proper health is maintained and are a healthy part of the human microbiome; However, disturbances to the local or systemic environment can lead to opportunistic infections such as periodontitis, gingivitis, or cavities .

It has been known that dental plaque plays a critical role in the development and progression of periodontal disease, gingivitis, and dental caries. Plaque control is the first line of defense against periodontal disease and gingival inflammation, and chemical plaque control methods should always be used in conjunction with mechanical methods .

Plaque removal is constantly maintained by mechanical techniques like toothbrushing and flossing, which are essential for controlling and preventing gingivitis, periodontitis, and dental caries. For mechanical plaque control, children need chemotherapeutic agents like therapeutic mouthwash since they lack the motivation or hand-eye coordination to reach the interproximal locations on their own.

Herbal medicine takes a preventative and promotional strategy. It is an integrated approach that treats diseases and promotes health by using a variety of treatments made from plants and their extracts. The use of natural herbs such as Triphala, Tulsi Patra, Jyestiamadh, Neem, Clove Oil, Pudina, Ajwain, and many more, either alone or in combination, has been shown by research to be a safe and effective treatment for a variety of oral health issues, including mouth ulcers, bleeding gums, halitosis, and tooth decay prevention .

Triphala, which exhibits antibacterial, antiseptic, and anti-inflammatory effects, is one of the most popular formulas in traditional Ayurvedic medicine. It is extensively used in dentistry and includes equal amounts of Terminalia Chebula, Terminalia Belerica, and Emblica Officinalis .

Triphala comprises tannins that facilitate the physical removal of microorganisms by aggregating them. This reduces the quantity of bacteria adhering to teeth during the initial phases of plaque development. Triphala mouth rinse exhibits extensive antibacterial activity against both Gram-positive and Gram-negative pathogens. It also demonstrates antioxidant properties that aid in minimizing dental plaque and gingivitis. The tannic acid in Triphala may facilitate plaque reduction by binding to bacterial cell surfaces that denature proteins and eradicate bacterial cells.

DETAILED DESCRIPTION:
The oral cavity possesses many kinds of bacterial communities. In a healthy condition, these bacteria are benign and represent a component of the human microbiome; however, changes in local or systemic environments can lead to opportunistic infections such as caries, gingivitis, or periodontitis (Vlam, 2019).

Gingivitis develops after 2 to 3 weeks of uninterrupted plaque accumulation, accompanied by a transition in subgingival bacteria from gram-positive to gram-negative species. Plaque-induced gingivitis, the most common form of periodontal disease, has been demonstrated by epidemiological studies to be frequent among dentate populations of all ages (Murakami et al., 2018; Deus and Ouanounou, 2022). In children aged 6 to 11, gingivitis was present in almost 73% of cases in developed nations. Besides, 50 - 99% of people develop gingivitis throughout adolescence (Pari et al., 2014).

Chlorhexidine (CHX) has established a reputation as the gold standard in chemical plaque reduction; however, long-term usage of CHX may result in a variety of problems, including dry mouth, changed taste perception, metallic taste, and tooth discoloration. Despite its anti-plaque capabilities, 0.12% CHX mouthwash has been associated with increased calculus deposition (Zanatta et al., 2010; Dandekar and Winnier, 2020). Thus, the quest for an ideal mouthwash with the beneficial properties of CHX without its side effects continues.

Triphala is one of the most popular formulations in ancient Ayurvedic medicine because it possesses antibacterial, antiseptic, and anti-inflammatory properties. It contains equal quantities of Terminalia Chebula, Terminalia Belerica, and Emblica Officinalis; it is commonly used in dentistry. Triphala was chemically examined and was discovered to have tannic acid, chebulic acid, and flavonoids as major ingredients (Minervini et al., 2024; Singaraju et al., 2024).

Triphala includes tannins, which assist in physically eliminating microorganisms by aggregating them together. This reduces the quantity of germs that attach to teeth during the initial stages of plaque development. Triphala mouth rinse has wide antibacterial properties against both Gram-positive and Gram-negative pathogens. It also has antioxidant properties that aid in reducing dental plaque and gingivitis (Minervini et al., 2024; Singaraju et al., 2024).

Numerous research studies have been done on the beneficial effects of Triphala mouthwashes on the management of plaque and gingivitis in adults. A knowledge gap persists regarding the effectiveness of Triphala mouthwash as an anti-plaque and anti-gingivitis among children and adolescents (Minervini et al., 2024).

Benefits of the study to participants:

* Provide a natural, effective herbal Mouthwash that provides antiplaque and anti-gingivitis properties.
* Minimal side effects.
* It will be cost-effective for the patient.

Benefits of the study to the community:

* Introducing a new mouthwash with minimal side effects.
* Improving the standards of pediatric dental care.
* Enhance the overall health of participants.

Benefits of the study for clinicians:

* Providing a new and alternative treatment option.
* Providing treatment with minimal side effects.
* Can be prescribed for a longer duration without fear of side effects. Explanation regarding the choice of comparators Chlorhexidine has been recommended as the gold standard for the treatment of gingivitis owing to its high success rate in the management of plaque accumulation and gingivitis when compared to other mouthwashes due to its antimicrobial and anti-inflammatory properties (Sharma et al., 2014).

Study Setting and Location

* Source of patients: This study will be conducted in the outpatient clinics of the Pediatric Dentistry and Dental Public Health Department - Faculty of Dentistry, Cairo University, Egypt.
* Operator: The Principal Investigator.
* Dental units: Knight Midmark Biltmore dental unit (Midmark Corporation 1700 S. Patterson Blvd., Suite 400, Dayton, Ohio 45409, USA).
* Instruments: Dental light, Mouth mirror & Periodontal probe.

The principal investigator will perform all clinical procedures as follows:

* Preoperative diagnostic procedures:

  1. Diagnostic charts with personal, medical, and dental history will be taken and recorded in the patient's diagnostic chart
  2. A clinical examination will be performed using a sterile mirror and probe to assess the eligibility criteria.
  3. if the patient fulfills the inclusion criteria, written informed consent will be obtained from the parents or the legal guardians, and verbal assent from the participant
  4. Preoperative and postoperative photographs will be taken.
  5. Baseline data, including both the gingival and plaque index, will be recorded in the patient diagnostic chart .
  6. Participants will be given meticulous oral hygiene instructions and appropriate brushing techniques.
  7. Patients will be allocated to the interventional or control groups with an allocation ratio 1: 1. Group I (Interventional group): Triphala mouthwash. Group II (Control group): Chlorhexidine mouthwash.

     For the interventional group (Triphala mouthwash):

     Participants will be supplied with 100 ml of prepared 6% Triphala mouthwash. They will be instructed to administer 15 ml of the mouthwash and swish it for 30 seconds two times daily under the supervision of their parents, 30 to 45 minutes after toothbrushing for 2 weeks. They will be instructed not to rinse or eat anything for 30 minutes after mouthwash use.

     Method of preparation of Triphala mouthwash:

     Triphala is available in a finely sieved powder form where a 6% Triphala mouthwash will be prepared according to (Bhattacharjee et al., 2015; Pradeep et al., 2016). Sixty grams (60 g) of pure Triphala powder will be dissolved in one liter of distilled water to obtain 6% of the extract. To improve patient compliance, two ml of glycerin will be added as a sweetening agent, and one ml of Pudin Hara will be added as a flavoring agent. The solution will be brought to boil for 10 minutes, then cooled and filtered. This mouthwash will be placed in opaque, sterile, sealed bottles.

     For the Control group (Chlorhexidine mouthwash):

     Participants will be supplied with 100 ml of commercially available 0.12% chlorhexidine mouthwash. About 10 ml will be administered, and participants will be asked to swish mouthwash for 30 seconds two times daily under the supervision of their parents, 30 to 45 minutes after toothbrushing for 2 weeks. They will be instructed not to rinse or eat anything for 30 minutes after mouthwash use.

     The strategies used to improve adherence to the intervention:

     The participants will be given a brushing calendar to mark every time they use mouthwash and bring this time at follow-up visits.

     Follow-up visits:

     The participants will be recalled after one week, two weeks, and three weeks.

     For outcome assessment:

     Training the examiners to conduct the clinical trial by the supervisors before the study initiation. The sessions will be conducted over two days. The first day will be an alignment session where the research team will review the clinical parameters in detail. The second day will be the assessment session when the principal investigator asses the patients with the characteristics of the study and the supervisors will evaluate the reliability of the examiner assessment.

     Primary outcome Plaque index :

     The Plaque index will be recorded using the mirror, periodontal probe, and disclosing agent to detect areas of plaque accumulation that will be stained by the disclosing agent at four areas for each tooth, including buccal, lingual, mesial, and distal.

     Criteria of plaque index:

  0 = No plaque.
  1. = Film of plaque adhering to the free gingival margin and adjacent area of the tooth.
  2. = Moderate accumulation of plaque within the gingival pocket.
  3. = An Abundance amount of plaque within the gingival pocket.

     To obtain the plaque index score for each tooth:

     The sum of the four tooth surface scores will be divided by four.

     Secondary outcome Gingival index:

     The gingival index will be recorded using a mirror and periodontal probe to assess the gingival status in four areas for each tooth, including buccal, lingual, mesial, and distal.

     Criteria of the gingival index:

  0 = Normal gingiva, no bleeding on probing & no inflammation.
  1. = Slight change in color & slight edema of the gingiva, mild inflammation, and no bleeding on probing.
  2. = Redness, edema, and glazing of the gingiva, moderate inflammation, and bleeding on probing.
  3. =Marked redness, edema, ulceration of the gingiva, severe inflammation, and spontaneous bleeding.

     To obtain the gingival index score for each tooth:

     The sum of the four tooth surface scores will be divided by four

     Sample size calculation:

     In a previous study by Shetty et al in 2021, the plaque index within the chlorohexidine group was normally distributed with a standard deviation of 0.94 after 21 days. If the true difference between the two groups is 1, we will need to study 15 children per group to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.8. The Type I error probability associated with this test of the null hypothesis is 0.05. The sample size was increased by 20% to compensate for possible dropouts to reach 18 children per group. Sample size was calculated using PS Power and Sample for Windows version 3.1.6 using an independent t-test.

     Recruitment and Recruitment Strategy:

     Patients attending the outpatient clinic of the Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University, Egypt, will be screened by the principal investigator until the target population is achieved. The patients will be subjected to a full examination and diagnosis using dental charts. Once the patients who are potentially eligible for this study are identified, they will be contacted by the principal investigator, who will explain the study and ascertain the patient's interest. If interested, more detailed evaluations and preparations will be made.

     Assignment of interventions

     Allocation:

     Random sequence Generation:

     The assistant supervisor will generate a random sequence using http://www.random.org/.

     Allocation Concealment Mechanism:

     The assistant supervisor will write the assigned group on a four-folded white paper and place it in a closed white envelope.

     Implementation:

     The participant will draw an envelope offered by the clinic nurse, and the patient's name will be written on it.

     Blinding:

     The trial participants, outcome assessors, and statisticians will be blinded.

     Bias:
* Selection bias will be avoided by randomization and allocation concealment.
* Performance bias will be overcome by performing all the procedures by the same principal investigator in a standardized way for all patients and blinding participants.
* Detection bias will be avoided by blinding the outcome assessor and detecting all study outcomes.
* Attrition bias will be avoided by understanding the reasons participants leave the study.
* Reporting bias will be avoided by registration of trials before the collection of data and reporting all study outcomes.

Baseline data collection:

Baseline data collection plans for assessment and collection of outcomes will be at 2 weeks and 3 weeks clinically by visual examination using a mirror and probe, and will be performed by two blinded assessors independently, and differences will be solved by consensus. To promote the quality of data, duplicate measurements by the same examiner (intra-examiner agreement) and training of assessors (inter-examiner agreement) will be done.

Data management:

The data will be entered into and stored on a personal computer. Another copy of the data will be saved on an external hard disc to prevent its loss.

Statistical analysis:

Data will be analyzed using Medcalc software, version 22 for Windows (MedCalc Software Ltd, Ostend, Belgium). Data will be explored for normality using the Kolmogorov-Smirnov test and the Shapiro-Wilk test. Continuous data will be described using mean and standard deviation. Intergroup comparison will be performed using the independent t-test, and intragroup comparison will be performed using repeated measures ANOVA, followed by Bonferroni-corrected pairwise comparisons. A P-value less than or equal to 0.05 will be considered statistically significant, and all tests will be two-tailed.

Monitoring :

The supervisors will frequently monitor the study's results, having complete access to the interim results, and will make the ultimate decision about the termination of the trial.

Harms:

* If there is an allergic reaction to mouthwash, stop it immediately and give the patient an antihistaminic drug.
* If staining is caused by chlorhexidine mouthwash, stop the mouthwash immediately and make polishing to the patient.
* If the Triphala mouthwash doesn't resolve the gingivitis, give the gold-standard mouthwash treatment.

Auditing:

The trial procedure and documentation will be regularly assessed by study supervisors. They will be involved in participant enrolment, consent, eligibility, and allocation to study groups; adherence to trial interventions and policies to protect participants, including reporting of complications and their treatments. They will supervise the performance of clinical procedures.

Research ethics approval :

This protocol, the template, and specific informed consent forms (local language and English versions) will be reviewed, approved, and agreed upon by the Research Ethics Committee will review all the nature of the interventions and will have the right to modify the study methods.

Protocol amendments :

The Ethics Committee will be notified of any administrative changes or modifications to the protocol. Any required changes during the trial period for the patient's interest that might affect the conduct of the study, including changes in the study objectives, study design, patient population, sample sizes, and intervention procedures, will require a formal amendment to the protocol. Such an amendment will be agreed upon by the Council of the Department of Pediatric Dentistry, Faculty of Dentistry, Cairo University.

Informed consent:

The investigator will discuss the trial with the legal guardian of each participating child:

* Verbal assents will be taken orally from the participants.
* Written informed consent will be taken from the legal guardian of each participant willing to participate in the trial. The consent form will be written in Arabic.

Confidentiality :

All data, information, participants' personal information, family history, and social and medical history will be stored in the files assigned to each patient with limited access to a minimum number of individuals necessary for quality control, audit, and analysis.

Declaration of interest :

This study is a part of a master's degree in Pediatric Dentistry, Faculty of Dentistry, Cairo University. No financial conflict of interest is confirmed. The study is self-funded by the principal investigator.

Access to data:

The investigator will be given access to data sets. All data sets will be password-protected. To ensure confidentiality, data dispersed to project team members will be blinded to any identifying participant information.

Post-trial care :

The investigator will offer full-mouth treatment, post-operative care, and preventive measures to all participants.

Dissemination policy:

The Thesis defense will be done as the study is a part of the requirements for a master's degree in Pediatric Dentistry.

Biological specimens:

There is no collection, laboratory evaluation, or storage of biological specimens in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 9 to 13 years.
* Apparently in good general health.
* Both sexes.
* Informed consent from their parents.
* Patients with fair oral hygiene and gingival inflammation.
* Participants should not have used mouthwashes for the follow-up period.

Exclusion Criteria:

* Patients with known allergies to any ingredient used in the study.
* History of immunosuppressive diseases.
* History of antibiotic or anti-inflammatory therapy in the previous month till the start of the study.
* Patients with orthodontic appliances.
* Parents refused to participate or were unable to attend follow-up visits.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The amount of plaque accumulation by using Plaque Index The plaque index will be recorded using the mirror, periodontal probe, and disclosing agent to detect areas of plaque accumulation that will be stained by the disclosing agent at tooth surfaces | From intervention till 3 weeks
  Criteria of plaque index:
  0 = No plaque.
  1. = Film of plaque adhering to the free gingival margin and adjacent area of the tooth.
  2. = Moderate accumulation of plaque within the gingival pocket.
  3. = An Abundance amount of plaque within the gingival pocket.
  To obtain the plaque index score for each tooth:
  The sum of the four tooth surface scores will be divided by four.

SECONDARY OUTCOMES:
Gingival health by using Gingival Index The gingival index will be recorded using a mirror and periodontal probe to assess the gingival status in four areas for each tooth including buccal, lingual, mesial, and distal. | From intervention till 3 weeks
  Criteria of the gingival index:
  0 = Normal gingiva, no bleeding on probing & no inflammation.
  1. = Slight change in color & slight edema of the gingiva, mild inflammation, and no bleeding on probing.
  2. = Redness, edema, and glazing of the gingiva, moderate inflammation, and bleeding on probing.
  3. =Marked redness, edema, ulceration of the gingiva, severe inflammation, and spontaneous bleeding.
  To obtain the gingival index score for each tooth:
  The sum of the four tooth surface scores will be divided by four.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Mohsen Aly, Study Chair — Finalizing the study design, revising the protocol, helping with the methodology, solving the existing problems, and revising the final version of the thesis.
Locations (1):
- Faculty of Dentistry Cairo Universty, Cairo, Egypt

REFERENCES:
- [Background] Zanatta FB, Antoniazzi RP, Rosing CK. Staining and calculus formation after 0.12% chlorhexidine rinses in plaque-free and plaque covered surfaces: a randomized trial. J Appl Oral Sci. 2010 Sep-Oct;18(5):515-21. doi: 10.1590/s1678-77572010000500015. PMID 21085810
- [Background] Van der Weijden FA, Van der Sluijs E, Ciancio SG, Slot DE. Can Chemical Mouthwash Agents Achieve Plaque/Gingivitis Control? Dent Clin North Am. 2015 Oct;59(4):799-829. doi: 10.1016/j.cden.2015.06.002. PMID 26427569
- [Background] Singaraju A, Nuvvula S, Rudravaram VR, Anchala K, Venkata Saikiran K, Mallineni SK. Efficacy of Triphala and Chlorhexidine Mouthwashes on Gingival Inflammation and Dental Plaque in Children: A Systematic Review. Oral. 2024 Nov 18;4(4):567-77.
- [Background] Shetty, Vabitha, Srikala Bhandary, and Roleen Pereira. "Evaluation of antiplaque and antimicrobial activity of Cocoa Bean Extract: An in vivo study." World 12.2 (2021): 151.
- [Background] Sharma A, Bansal P, Grover A, Sharma S, Sharma A. Oral health status and treatment needs among primary school going children in Nagrota Bagwan block of Kangra, Himachal Pradesh. J Indian Soc Periodontol. 2014 Nov-Dec;18(6):762-6. doi: 10.4103/0972-124X.147421. PMID 25624634
- [Background] Bhattacharjee R, Nekkanti S, Kumar NG, Kapuria K, Acharya S, Pentapati KC. Efficacy of triphala mouth rinse (aqueous extracts) on dental plaque and gingivitis in children. J Investig Clin Dent. 2015 Aug;6(3):206-10. doi: 10.1111/jicd.12094. Epub 2014 May 22. PMID 24850703
- [Background] Minervini G, Marrapodi MM, Tirupathi S, Afnan L, Di Blasio M, Cervino G, Isola G, Cicciu M. Comparative anti-plaque and anti-gingivitis efficiency of Triphala versus chlorhexidine mouthwashes in children: a systematic review and meta-analysis. J Clin Pediatr Dent. 2024 Sep;48(5):51-59. doi: 10.22514/jocpd.2024.103. Epub 2024 Sep 3. PMID 39275820
- [Background] Fan W, Liu C, Zhang Y, Yang Z, Li J, Huang S. Epidemiology and associated factors of gingivitis in adolescents in Guangdong Province, Southern China: a cross-sectional study. BMC Oral Health. 2021 Jun 16;21(1):311. doi: 10.1186/s12903-021-01666-1. PMID 34134691
- [Background] Fahim MFM, Zarnigar P. Effect of prepared herbal mouthwash in maintaining the oral health of school children: A single-blind randomised control trial. Explore (NY). 2024 Jul-Aug;20(4):535-543. doi: 10.1016/j.explore.2023.12.003. Epub 2023 Dec 15. PMID 38594113
- [Background] Poppolo Deus F, Ouanounou A. Chlorhexidine in Dentistry: Pharmacology, Uses, and Adverse Effects. Int Dent J. 2022 Jun;72(3):269-277. doi: 10.1016/j.identj.2022.01.005. Epub 2022 Mar 12. PMID 35287956
- [Background] Chrysanthakopoulos, N. A. (2016). Prevalence of gingivitis and associated factors in 13-16-year-old adolescents in Greece. European Journal of General Dentistry, 5(02), 58-64
- [Background] Bhat N, Mitra R, Oza S, Mantu VK, Bishnoi S, Gohil M, Gupta R. The antiplaque effect of herbal mouthwash in comparison to chlorhexidine in human gingival disease: a randomized placebo controlled clinical trial. J Complement Integr Med. 2014 Jun;11(2):129-37. doi: 10.1515/jcim-2014-0002. PMID 24698829
- [Background] 3. Bhat, N., Ruchi Mitra, R. M., Reddy, J. J., Swapnil Oza, S. O., & Vinayak, K. M. (2013). Evaluation of efficacy of chlorhexidine and a herbal mouthwash on dental plaque: an in vitro comparative study
- [Background] Barnett ML. The role of therapeutic antimicrobial mouthrinses in clinical practice: control of supragingival plaque and gingivitis. J Am Dent Assoc. 2003 Jun;134(6):699-704. doi: 10.14219/jada.archive.2003.0255. PMID 12839405
- [Background] Pari A, Ilango P, Subbareddy V, Katamreddy V, Parthasarthy H. Gingival diseases in childhood - a review. J Clin Diagn Res. 2014 Oct;8(10):ZE01-4. doi: 10.7860/JCDR/2014/9004.4957. Epub 2014 Oct 20. PMID 25478471
- [Background] Dandekar NV, Winnier JJ. Assessment of Antiplaque and Anti-Gingivitis Efficacy of Mouthwashes Prepared from Neem and Mango Extracts. Front Dent. 2020 Jun 20;17:11. doi: 10.18502/fid.v17i11.4128. eCollection 2020. PMID 35968157
- [Background] Bajaj N, Tandon S. The effect of Triphala and Chlorhexidine mouthwash on dental plaque, gingival inflammation, and microbial growth. Int J Ayurveda Res. 2011 Jan;2(1):29-36. doi: 10.4103/0974-7788.83188. PMID 21897640